CLINICAL TRIAL: NCT00346840
Title: Controlled-Release Misoprostol Vaginal Insert in Parous Women for Labor Induction: Randomized Trial
Brief Title: Safety and Efficacy Study of Misoprostol Vaginal Insert for Induction of Labour
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Miso-Obs-002
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Labor Induction; Cervical Ripening
Keywords: Labor induction; cervical ripening; misoprostol; vaginal insert

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MVI 25 (Experimental): Misoprostol vaginal insert 25 mcg
  Interventions: Drug: Misoprostol vaginal insert 25 mcg
- MVI 50 (Experimental): Misoprostol vaginal insert 50 mcg
  Interventions: Drug: Misoprostol vaginal insert 50 mcg
- MVI 100 (Experimental): Misoprostol vaginal insert 100 mcg
  Interventions: Drug: Misoprostol vaginal insert 100 mcg
- MVI 200 (Experimental): Misoprostol vaginal insert 200 mcg
  Interventions: Drug: Misoprostol vaginal insert 200 mcg

INTERVENTIONS:
Drug: Misoprostol vaginal insert 25 mcg — One hydrogel polymer vaginal insert for up to 24h
  Other Names: Misoprostol vaginal insert
  Arms: MVI 25
Drug: Misoprostol vaginal insert 50 mcg — One hydrogel polymer vaginal insert for up to 24h
  Other Names: Misoprostol vaginal insert
  Arms: MVI 50
Drug: Misoprostol vaginal insert 100 mcg — One hydrogel polymer vaginal insert for up to 24h
  Other Names: Misoprostol vaginal insert
  Arms: MVI 100
Drug: Misoprostol vaginal insert 200 mcg — One hydrogel polymer vaginal insert for up to 24h
  Other Names: Misoprostol vaginal insert
  Arms: MVI 200

SUMMARY:
The primary objective of the study was assessment of the efficacy of four dose reservoirs (25 mcg, 50 mcg, 100 mcg, 200 mcg) of intravaginal controlled release misoprostol administered for up to 24 hours. Efficacy was measured in terms of time from insert placement to vaginal delivery.

DETAILED DESCRIPTION:
Approximately 20% of pregnant women require medical intervention to induce labour for reasons including post-date pregnancy, pre-eclampsia, maternal diabetes, premature rupture of the membranes and intra-uterine fetal growth retardation. There are two fundamental changes that characterise pre-labour preparation for delivery: sensitisation of the myometrium to produce contractions, and ripening (softening and dilation) of the cervix. Prostaglandins (PG) are fundamental to both of these changes, and several forms have been used to successfully induce labour. Dinoprostone (PGE2) is an example of a cervical ripening agent that is available in gel and tablet form and has a proven record of successful cervical ripening in this population. Dinoprostone is also available in a controlled release vaginal delivery system, which is manufactured by Controlled Therapeutics (Scotland) a subsidiary of Cytokine PharmaSciences, Inc., King of Prussia, PA, USA.

Another synthetic prostaglandin that has been shown to be an effective cervical ripener and labour inducer is misoprostol. Oral tablets are broken into fragments and used intravaginally to ripen the cervix and induce labour Due to the disadvantages of existing cervical ripeners (delivery of bolus doses, freezer or refrigerated storage, lack of efficacy in labour induction), and due to safety concerns with the off-label use of oral misoprostol tablet fragments, Controlled Therapeutics has developed a controlled release vaginal delivery system similar to its marketed dinoprostone product but containing misoprostol.

This study examines four dose strengths of the misoprostol vaginal insert in women who need to have their labours induced.

ELIGIBILITY:
Inclusion Criteria:

* At term (37 to 42 weeks inclusive gestation).
* Aged 18 years or older.
* One previous full term delivery (at least 37 weeks gestation).
* Singleton pregnancy.
* Cephalic presentation (normal lie).
* Bishop score more than 6 as determined by MBS criteria.
* Uncomplicated pregnancy as judged by the physician.
* Written informed consent.

Exclusion Criteria:

* four previous full term deliveries.
* Previous uterine surgery, including C-section and surgery to the cervix of the uterus (cone biopsy of the cervix is permitted).
* In spontaneous labour.
* Administration of oxytocin or a tocolytic drug or any other cervical ripening or labour inducing agent prior to enrolment (within seven days of enrolment).
* Suspected cephalo-pelvic disproportion.
* Evidence or suggestion of fetal distress.
* Subject has received NSAID (including aspirin) within four hours of study treatment (topical is permitted).
* Pyrexia (oral or aural temperature > 37.5C).
* Unexplained genital bleeding during this pregnancy after 24 weeks.
* Current pelvic inflammatory disease, unless adequate prior treatment has been instituted.
* Placenta praevia.
* Known or suspected allergy to misoprostol or other prostaglandins.
* Prior serious adverse event related to prostaglandin administered by any route for any indication.
* Subject unable to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2003-06; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Time to vaginal delivery. | From insertion of study drug to neonate delivery

SECONDARY OUTCOMES:
uterine hyperstimulation | From insertion of study drug to neonate delivery
safety in terms of maternal, fetal and neonatal adverse events | From insertion of study drug to neonate delivery
Success on composite modified Bishop score (MBS)at 12 hours after drug insertion | From insertion of study drug to 12 hours
frequency and amount of oxytocin use | From insertion of study drug to neonate delivery
drug release characteristics in terms of residual concentrations | From insertion of study drug to removal of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Pleiad, Inc.
Locations (6):
- United Kingdom (6):
  - Birmingham Women's Hospital, Birmingham
  - Princess Royal Maternity Hospital, Glasgow
  - King George Hospital, Ilford
  - Liverpool Women's Hospital, Liverpool
  - Northampton General Hospital, Northampton
  - The Queen's Mother's Hospital, Yorkhill, Glasgow

REFERENCES:
- [Background] Castaneda CS, Izquierdo Puente JC, Leon Ochoa RA, Plasse TF, Powers BL, Rayburn WF. Misoprostol dose selection in a controlled-release vaginal insert for induction of labor in nulliparous women. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 2):1071-5. doi: 10.1016/j.ajog.2005.06.072. PMID 16157114
- [Background] Rayburn WF, Powers BL, Plasse TF, Carr D, Di Spirito M. Pharmacokinetics of a controlled-release misoprostol vaginal insert at term. J Soc Gynecol Investig. 2006 Feb;13(2):112-7. doi: 10.1016/j.jsgi.2005.10.004. PMID 16443504
- [Result] Ewert K, Powers B, Robertson S, Alfirevic Z. Controlled-release misoprostol vaginal insert in parous women for labor induction: a randomized controlled trial. Obstet Gynecol. 2006 Nov;108(5):1130-7. doi: 10.1097/01.AOG.0000239100.16166.5a. PMID 17077234